CLINICAL TRIAL: NCT07115303
Title: Results of Laparoscopic Appendectomy With Application of Clips Versus Ligature for Stump Closure: A Comparative Study
Brief Title: Results of Laparoscopic Appendectomy With Application of Clips Versus Ligature for Stump Closure
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Ahmed Amer Abdelraheem, Resident of General, Oncologic& Laparscopic Surgery Faculty of Medicine, Sohag University, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med-25-7---18MS
Record Dates: First submitted 2025-08-04; First posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Appendicitis
MeSH Terms: conditions — Appendicitis | interventions — Ligation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laparoscopic Appendectomy with application of clips for stump closure (Active Comparator)
  Interventions: Procedure: Laparoscopic Appendectomy with application of clips for stump closure
- Laparoscopic Appendectomy with ligature for stump closure (Active Comparator)
  Interventions: Procedure: Laparoscopic Appendectomy with ligature for stump closure

INTERVENTIONS:
Procedure: Laparoscopic Appendectomy with application of clips for stump closure — in patients who will undergo Laparoscopic Appendectomy, appendicular stump will be closed by application of clips
  Arms: Laparoscopic Appendectomy with application of clips for stump closure
Procedure: Laparoscopic Appendectomy with ligature for stump closure — in patients who will undergo Laparoscopic Appendectomy, appendicular stump will be closed by ligation
  Arms: Laparoscopic Appendectomy with ligature for stump closure

SUMMARY:
This a prospective study to compare between clipping and ligation of appendicular stump in laparoscopic appendectomies regarding ;technical feasibility , post operative complications as fecal fistula and economic consideration.

ELIGIBILITY:
Inclusion Criteria:

* Any patient diagnosed with acute appendicitis of any age and of any sex presented to ER of the Department of General, Laparoscopic and Oncologic Surgery Department, Sohag University Hospital will be enrolled in this study.

Exclusion Criteria:

* Patients with complicated appendicitis.
* Patients with unstable cardiac or pulmonary condition.
* Patients with suspicious crhon's disease or mass intraoperative.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-07-14 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Results of Laparoscopic Appendectomy with application of clips versus ligature for stump closure | 24 hours postoperative
  postoperative hospital stay

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university hospital, Sohag, Egypt

REFERENCES:
- [Background] Makaram N, Knight SR, Ibrahim A, Patil P, Wilson MSJ. Closure of the appendiceal stump in laparoscopic appendectomy: A systematic review of the literature. Ann Med Surg (Lond). 2020 Aug 4;57:228-235. doi: 10.1016/j.amsu.2020.07.058. eCollection 2020 Sep. PMID 32802324
- [Background] Farahani PK, Safaei N. Comparison of two methods: Clipping and suturing in laparoscopic appendectomy. Surg Open Sci. 2024 May 3;19:162-165. doi: 10.1016/j.sopen.2024.04.007. eCollection 2024 Jun. PMID 38764557
- [Background] Poon SHT, Law SY, Lai ATY. Clips closure versus endoloop ligation in laparoscopic appendectomy: a systematic review and meta-analysis of comparative studies. Ann Med Surg (Lond). 2023 Sep 6;85(10):5011-5021. doi: 10.1097/MS9.0000000000001260. eCollection 2023 Oct. PMID 37811063